CLINICAL TRIAL: NCT00013104
Title: Implementation of Ischemic Heart Disease Clinical Practice Guidelines
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: VCR 99-014
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-01

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this study is to design and evaluate targeted implementation strategies to fully integrate the VHA clinical practice guidelines for ischemic heart disease into VHA clinical practice. Effectively implementing the guideline will enhance the quality, appropriateness, timeliness, and cost effectiveness of care delivered to veterans with ischemic heart disease.

DETAILED DESCRIPTION:
Background:

The purpose of this study is to design and evaluate targeted implementation strategies to fully integrate the VHA clinical practice guidelines for ischemic heart disease into VHA clinical practice. Effectively implementing the guideline will enhance the quality, appropriateness, timeliness, and cost effectiveness of care delivered to veterans with ischemic heart disease.

Objectives:

The long-term objective of this study is to identify the best strategies for implementing the IHD guidelines to improve guideline adherence and provider acceptance. The specific objectives of the study are to: 1) describe the temporal aspects of guideline acceptance and adherence over three periods of time: pre-implementation, post-implementation of general strategies, and post- implementation of targeted strategies; 2) assess the relative effectiveness of targeted intervention strategies on guideline adherence; 3) identify the relationships among provider beliefs, attitudes, and their intentions to use guidelines; 4) identify the costs associated with implementation of general and targeted implementation strategies; and 5) describe provider satisfaction with targeted implementation strategies.

Methods:

Qualitative (focus groups, interviews with key informants) and quantitative methods (surveys, chart reviews) are used to address study objectives. A survey will be sent to providers to measure beliefs and attitudes that predict provider acceptance to clinical practice guidelines. Patient level data will be collected from reviews of charts from each facility. Based on provider focus groups we will design targeted strategies to overcome system barriers and address needs identified by providers to support clinical practice guideline implementation. A randomized trial will be conducted to assess the relative effectiveness of the targeted intervention strategies.

Status:

Data collection has ended. We are currently evaluating adherence data at all sites following introduction of case management to determine if the intervention increases adherence to the guidelines.

ELIGIBILITY:
Inclusion Criteria:

None

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L. Nelson, RN PhD FAAN, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States